CLINICAL TRIAL: NCT02154360
Title: A Phase IB, Open Label Study to Examine the Safety, Pharmacokinetic Characteristics and Anti-Inflammatory Effects of the NK-1R Antagonist, Aprepitant, In HIV-Infected Subjects Receiving Atazanavir/Ritonavir Or Darunavir/Ritonavir
Brief Title: Pharmacokinetic Characteristics and Anti-Inflammatory Effects of Aprepitant In HIV-Infected Subjects
Acronym: Emend-IV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPenn 819693
Record Dates: First submitted 2014-05-22; First posted 2014-06-03 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: HIV Infection
Keywords: HIV infection; NK-1R antagonists; aprepitant; ritonavir boosting
MeSH Terms: conditions — HIV Infections | interventions — Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aprepitant (Experimental): Subjects will add 375 mg daily dosing of aprepitant (Emend®) to their current antiretroviral therapy for 28 days.
  * 6 participants will be receiving an antiretroviral regimen containing atazanavir/ritonavir (300/100 mg) daily plus two other antiretrovirals.
  * 6 participants will be receiving an antiretroviral regimen containing darunavir/ritonavir (800/100 mg) daily plus two other antiretrovirals.
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant — Subjects will add 375 mg daily dosing of aprepitant (Emend®) to their current antiretroviral therapy for 28 days
  Other Names: Emend

SUMMARY:
This is an open-label, single arm, phase I study to determine the safety, PK characteristics and anti-inflammatory effects of the NK-R1 coadministered with ritonavir-containing antiretroviral therapy in individuals with well-controlled viral replication.

Our hypothesis is that Aprepitant will be safe, well tolerated, and will have anti-inflammatory properties when administered concomitantly with the protease inhibitor ritonavir.

DETAILED DESCRIPTION:
This is an open-label, single arm, phase I study to determine the safety, PK characteristics and anti-inflammatory effects of the NK-R1 coadministered with ritonavir-containing antiretroviral therapy in individuals with well-controlled viral replication.

Our hypothesis is that Aprepitant will be safe, well tolerated, and will have anti-inflammatory properties when administered concomitantly with the protease inhibitor ritonavir. The study will recruit 12 participants receiving either darunavir/ritonavir or atazanavir/ritonavir

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
2. Antiretroviral treatment with a regimen that includes either atazanavir 300 mg daily with ritonavir 100 mg daily or darunavir/ritonavir on a combination of 800/100 mg daily for at least 6 months prior to enrollment.
3. CD4+ cell count ≥ 350/mm3 for at least 6 months prior to enrollment and performed at any CLIA-certified laboratory.
4. Plasma HIV-1 RNA below the limit of quantification of an ultrasensitive assay as measured by any standard assay (the Roche Amplicor, the UltraSensitive HIV-1 Monitor assay (Roche Molecular Systems), or Version 3 bDNA assay or other) for at least 6 months prior to enrollment by any laboratory that is CLIA-certified (or its equivalent) for the assay.
5. Laboratory values obtained within 30 days prior to study entry, as follows:

   * Absolute neutrophil count (ANC) greater or equal than 750/mm3
   * Hemoglobin greater or equal than 10.0 g/dL
   * Platelet count greater or equal than 100,000/mm3
   * Creatinine less or equal than 2 x ULN (fasting)
   * AST (SGOT), ALT (SGPT), and alkaline phosphatase less or equal than 2 x ULN
   * Total bilirubin less or equal than 2.5 x ULN
   * Albumin greater or equal than 3 g/dL
6. Female subjects of reproductive potential must have a negative spot urine pregnancy test result (with a sensitivity of at least 50 mIU/mL) performed at entry, prior to starting initial study treatment.
7. All subjects must agree not to participate in a conception process while on study drug and for 30 days after stopping the medication.

   If participating in sexual activity that could lead to pregnancy, the female study subject must use at least one of the forms of contraception listed below while receiving the protocol-specified medication and for 30 days after stopping the medication.
   * Condoms (male or female) with or without a spermicidal agent
   * Diaphragm or cervical cap with spermicide
   * IUD

   Female subjects, who are not of reproductive potential defined as women who have been post-menopausal for at least 24 consecutive months, or women who have undergone surgical sterilization, (e.g. hysterectomy, bilateral oophorectomy, or salpingotomy) are eligible without requiring the use of contraception. Subject reported history is acceptable for documentation of sterilization, other contraceptive methods, menopause and a female's reproductive potential.
8. Karnofsky performance score greater or equal than 80 within 30 days prior to study entry (Appendix I).
9. Men and women greater or equal than 18 years of age.
10. Ability and willingness of subject or legal guardian/representative to give written informed consent.
11. Willing to return for a follow-up visit on day 58.
12. Subjects taking any precautionary concomitant medications must be on stable doses for >8 weeks prior to study entry and have no plans to change medications or doses for the duration of the study.

Exclusion Criteria:

1. Diabetes requiring treatment with oral hypoglycemics or insulin therapy.
2. Pregnancy within 90 days prior to study entry.
3. Use of inhibitors of metabolism by the cytochrome P450 3A4 with the exception of ritonavir, atazanavir and darunavir (i.e. Diltiazem, Ketoconazole, Clarithromycin, Nelfinavir, Itraconazole, Nefazodone, Troleandomycin)
4. Use of inducers of metabolism by the cytochrome P450 3A4 (i.e.: Rifampin, Carbamazepine, Phenytoin) with the exception of the protease inhibitors considered in this trial.
5. Breast-feeding.
6. Use of systemic corticosteroids or hormonal agents within 90 days prior to study entry.
7. Use of any immunomodulator, HIV vaccines, or investigational therapy within 90 days prior to study entry. However, if the experimental agent has a short half life, as determined by the Principal Investigator, the required wash out period can be reduced to 30 days.
8. Any vaccination within 30 days prior to study entry.
9. Use of systemic cytotoxic chemotherapy within 90 days prior to study entry.
10. History of allergy to aprepitant or its formulations.
11. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
12. History of chronic active hepatitis B or C infection or severe hepatic dysfunction (Child-Pugh score > 9) regardless of etiology
13. Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 14 days prior to study entry.
14. Weight < 40 kg or 88 lbs. within 90 days prior to study entry.
15. History of severe psychiatric comorbidities, such as depression, schizophrenia, mania, psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Inflammatory | 14 days
  Change in levels of Soluble CD163 from baseline to Day 14.
Safety | 28 days
  Incidence of Grade 2, 3, and 4 adverse events (using the DAIDS grading scale) by body system and by type. Lack of virologic control is considered a safety event for the purpose of this trial.
Pharmacokinetic Cmin: | day 1, 14 and 28
  Trough plasma aprepitant concentration.
Pharmacokinetic Cmax | day 1, 14 and 28
  Maximum plasma concentration.
Pharmacokinetic Tmax | day 1, 14 and 28
  Time to maximum plasma concentration
Pharmacokinetic AUCss | day 1, 14 and 28
  Area under the plasma concentration-time curve at steady-state (based on steady-state assessment of trough concentrations or via modeling).

SECONDARY OUTCOMES:
Inflammatory markers | 28 days
  * Change in levels of Soluble CD163 from baseline to Day 28 and 58
  * Plasma SP levels
  * CD4/PD-1 expression
Lipids | 28 days
  * Triglycerides
  * Total cholesterol
  * HDL
  * LDL
  * Insulin
Neurological | 28 days
  * Hamilton-17 Depression Rating Scale (HAM-D-17) score
  * Hamilton- Anxiety Symptoms (HAM-A) score
  * Pittsburgh Sleep Quality Index (PSQI) score

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania Clinical Research Site, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Tebas P, Tuluc F, Barrett JS, Wagner W, Kim D, Zhao H, Gonin R, Korelitz J, Douglas SD. A randomized, placebo controlled, double masked phase IB study evaluating the safety and antiviral activity of aprepitant, a neurokinin-1 receptor antagonist in HIV-1 infected adults. PLoS One. 2011;6(9):e24180. doi: 10.1371/journal.pone.0024180. Epub 2011 Sep 8. PMID 21931661
- [Background] Manak MM, Moshkoff DA, Nguyen LT, Meshki J, Tebas P, Tuluc F, Douglas SD. Anti-HIV-1 activity of the neurokinin-1 receptor antagonist aprepitant and synergistic interactions with other antiretrovirals. AIDS. 2010 Nov 27;24(18):2789-96. doi: 10.1097/QAD.0b013e3283405c33. PMID 20975512
- [Background] Wang X, Douglas SD, Lai JP, Tuluc F, Tebas P, Ho WZ. Neurokinin-1 receptor antagonist (aprepitant) inhibits drug-resistant HIV-1 infection of macrophages in vitro. J Neuroimmune Pharmacol. 2007 Mar;2(1):42-8. doi: 10.1007/s11481-006-9059-6. Epub 2007 Jan 12. PMID 18040825
- [Derived] Spitsin S, Tebas P, Barrett JS, Pappa V, Kim D, Taylor D, Evans DL, Douglas SD. Antiinflammatory effects of aprepitant coadministration with cART regimen containing ritonavir in HIV-infected adults. JCI Insight. 2017 Oct 5;2(19):e95893. doi: 10.1172/jci.insight.95893. PMID 28978797